CLINICAL TRIAL: NCT03311087
Title: Conduct of High Flow Nasal Cannula Oxygen During Acute Hypoxemic Respiratory Failure: a Multicentre Observational Study
Brief Title: Conduct of Nasal High Flow Oxygen in Acute Respiratory Failure
Acronym: DECIPHEROBS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hôpital Louis Mourier (Other)
Responsible Party: Principal Investigator, Prof Jean-Damien RICARD, Professor of Intensive Care Medicine, Hôpital Louis Mourier
Other Study IDs: HLM_JDR6
Record Dates: First submitted 2017-10-11; First posted 2017-10-16 (Actual); Last update posted 2018-07-20 (Actual); Status verified 2018-07

CONDITIONS: Acute Respiratory Failure With Hypoxia; Hypoxemia
Keywords: high flow nasal oxygen; acute hypoxemic respiratory failure; adults; intensive care unit
MeSH Terms: conditions — Hypoxia; Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Although many studies have investigated the clinical benefits of nasal high flow during acute hypoxemic respiratory failure, there is no data (and even less so recommendations) on how to best conduct this technique, including its initiation and its weaning periods. Investigators will assess in a multicenter, observational study, the way clinicians use nasal high flow therapy in patients with acute respiratory failure in order to try identify one or more strategies that may be then compared in an interventional study.

DETAILED DESCRIPTION:
Nasal high flow oxygen therapy is increasingly used as a first-line treatment for hypoxemic acute respiratory failure, because of its remarkable tolerance (in comparison with NIV) and its physiological effects (nasopharyngeal dead space washout, positive end-expiratory pressure effect with possible alveolar recruitment, better matching with the patient's inspiratory flow, more reliable and adjustable FiO2); that together contribute to a reduction in respiratory workload and better oxygenation.

Although many studies have investigated the clinical benefits of nasal high flow during acute hypoxemic respiratory failure, there are no data (and even less recommendations) on how to best conduct this technique, including its initiation and its weaning periods.

Because different approaches exist among clinicians, investigators believe that a multicenter observational study that would collect data regarding the different ways high flow is conducted in patients with acute respiratory failure is necessary before performing an interventional study that would test and compare different strategies in order to answer the question: what are the best strategies (in terms of flow and FiO2 settings) to initiate and to wean high-flow oxygen therapy in patients with acute respiratory failure?

Investigators will assess in a multicenter, observational study, the way clinicians use nasal high flow therapy in patients with acute respiratory failure in order to try identify one or more strategies that may be then compared in an interventional study.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 or older
* admitted to the intensive care unit (ICU) or to the intermediate care for acute hypoxemic respiratory failure (whatever the cause)
* treated with nasal high flow oxygen therapy
* with a minimal FiO2 of FiO2≥50% and a gas flow ≥40 L/min
* anticipated duration of nasal high flow therapy greater or equal to 24 hours

Non-inclusion Criteria:

* prophylactic, post-extubation nasal high flow therapy
* palliative nasal high flow therapy (do-not-resuscitate order)

Exclusion criteria

- nasal high flow therapy administered for less than 24 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted to an ICU or an intermediate care unit, who require nasal high flow oxygen therapy for acute hypoxemic respiratory failure
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-07-09 (Actual); Primary Completion 2018-10 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
values of gas flow over time (in liters per minute) | entire duration of high flow therapy (5 to 7 days)
  values of gas flow set on the device of nasal high flow will be monitored over time so as to describe how physicians set and modify this parameter during treatment with nasal high flow
values of fraction in inspired oxygen (FiO2) over time (between 0.21 and 1.0) | entire duration of high flow therapy (5 to 7 days)
  values of FiO2 set on the device of nasal high flow will be monitored over time so as to describe how physicians set and modify this parameter during treatment with nasal high flow

SECONDARY OUTCOMES:
respiratory rate (breath per minute) | entire duration of high flow therapy (5 to 7 days)
  values of respiratory rate upon initiation of nasal high flow and at each change of nasal high flow parameters (gas flow or FiO2) will be monitored.
pulse oximetry (SpO2) (percentage) | entire duration of high flow therapy (5 to 7 days)
  values of oxgen saturation upon initiation of nasal high flow and at each change of nasal high flow parameters (gas flow or FiO2) will be monitored.
values of the Respiratory rate Oxygenation indeX ("ROX") index defined as the ratio of pulse oximetry over fraction of inspired oxygen to respiratory rate | 12 hours
  values of the "ROX" index will be monitored at different time points (2, 6 and 12 hours after nasal high flow therapy initiation)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Damien Ricard, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (10):
- France (10):
  - Service de Réanimation Médico-Chirurgicale, Colombes
  - Service de Réanimation Médicale, Dijon
  - Service de Réanimation Médicale, Grenoble
  - Service de Réanimation, Longjumeau
  - Service de Réanimation, Orléans
  - Service de Réanimation Médicale et Resiratoire, Paris
  - Service de Réanimation Médicale, Paris
  - Service de Réanimation, Poitiers
  - Service de Réanimation Médicale, Rouen
  - Service de Réanimation Médicale, Tours

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Frat JP, Thille AW, Mercat A, Girault C, Ragot S, Perbet S, Prat G, Boulain T, Morawiec E, Cottereau A, Devaquet J, Nseir S, Razazi K, Mira JP, Argaud L, Chakarian JC, Ricard JD, Wittebole X, Chevalier S, Herbland A, Fartoukh M, Constantin JM, Tonnelier JM, Pierrot M, Mathonnet A, Beduneau G, Deletage-Metreau C, Richard JC, Brochard L, Robert R; FLORALI Study Group; REVA Network. High-flow oxygen through nasal cannula in acute hypoxemic respiratory failure. N Engl J Med. 2015 Jun 4;372(23):2185-96. doi: 10.1056/NEJMoa1503326. Epub 2015 May 17. PMID 25981908
- [Background] Sztrymf B, Messika J, Bertrand F, Hurel D, Leon R, Dreyfuss D, Ricard JD. Beneficial effects of humidified high flow nasal oxygen in critical care patients: a prospective pilot study. Intensive Care Med. 2011 Nov;37(11):1780-6. doi: 10.1007/s00134-011-2354-6. Epub 2011 Sep 27. PMID 21946925
- [Background] Sztrymf B, Messika J, Mayot T, Lenglet H, Dreyfuss D, Ricard JD. Impact of high-flow nasal cannula oxygen therapy on intensive care unit patients with acute respiratory failure: a prospective observational study. J Crit Care. 2012 Jun;27(3):324.e9-13. doi: 10.1016/j.jcrc.2011.07.075. Epub 2011 Sep 29. PMID 21958974
- [Background] Messika J, Ben Ahmed K, Gaudry S, Miguel-Montanes R, Rafat C, Sztrymf B, Dreyfuss D, Ricard JD. Use of High-Flow Nasal Cannula Oxygen Therapy in Subjects With ARDS: A 1-Year Observational Study. Respir Care. 2015 Feb;60(2):162-9. doi: 10.4187/respcare.03423. Epub 2014 Nov 4. PMID 25371400
- [Background] Roca O, Messika J, Caralt B, Garcia-de-Acilu M, Sztrymf B, Ricard JD, Masclans JR. Predicting success of high-flow nasal cannula in pneumonia patients with hypoxemic respiratory failure: The utility of the ROX index. J Crit Care. 2016 Oct;35:200-5. doi: 10.1016/j.jcrc.2016.05.022. Epub 2016 May 31. PMID 27481760